CLINICAL TRIAL: NCT04653103
Title: Prevalence of NASH in Subjects With Different Classes of Obesity
Brief Title: NASH in Subjects With Different Classes of Obesity
Acronym: CONNECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Professor, Catholic University of the Sacred Heart
Other Study IDs: 20202011
Record Dates: First submitted 2020-11-20; First posted 2020-12-04 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NAFLD; Obesity; Obesity, Morbid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with obesity: Subjects with different classes of obesity
  Interventions: Procedure: Liver biopsy

INTERVENTIONS:
Procedure: Liver biopsy — Biopsy of the liver to assess for Non-alcoholic steatohepatitis

SUMMARY:
It is an observational trial on 500 subjects. The purpose of this trial is to assess the prevalence of non-alcoholic steatohepatitis (NASH) in subjects with different classes of obesity.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is rapidly becoming the most common cause of chronic liver disease due to an increase in the prevalence of obesity. The development of NASH leads to an increase in morbidity and mortality. Since patients with obesity are at an increased risk of NASH, the aim of this trial is to assess the prevalence of NASH in this class of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 69 years

Exclusion Criteria:

* Pregnancy
* Active cancer
* End stage renal failure
* End stage liver failure
* Being unable to understand and sign informed consent

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with different classes of obesity
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NASH | 6 months
  Prevalence of NASH in a cohort of patients with different classes of obesity

SECONDARY OUTCOMES:
Assessment of lipid profile | 6 months
  Assessment of triglycerides, total cholesterol, LDL and HDL cholesterol
Assessment of glycemic profile | 6 months
  Assessment of fasting glucose
Assessment of glycated hemoglobin | 6 months
  Assessment of glycated hemoglobin
Assessment of liver enzymes | 6 months
  Assessment of AST, ALT, GGT
Assessment of insulin | 6 months
  Assessment of fasting insulin
Assessment of metabolic profile | 6 months
  Assessment of HOMA-IR index

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - University of Rome Sapienza, Roma
  - Catholic University School of Medicine, Rome

IPD SHARING:
Plan to Share IPD: No